CLINICAL TRIAL: NCT03666078
Title: Assessment of Maternal and Perinatal Morbidity and Mortality in Vaginal and Cesarean Delivery Among a Sample of Women Delivering at Ain Shams University Maternity Hospital
Brief Title: Assessment of Maternal and Perinatal Morbidity and Mortality in Vaginal and Cesarean Delivery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alzahraa Ismail Ragheb Goda (Other)
Responsible Party: Sponsor-Investigator, Alzahraa Ismail Ragheb Goda, resident of obstetrics and gynecology, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: zahra2018
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Delivery ,Complications,Maternal; Delivery,Complication,Fetal
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal vaginal delivery
- assisted vaginal delivery
- elective cesarean delivery
  Interventions: Procedure: cesarean delivery
- emergency cesarean delivery
  Interventions: Procedure: cesarean delivery

INTERVENTIONS:
Procedure: cesarean delivery — women delivered by cesarean section
  Groups: elective cesarean delivery; emergency cesarean delivery

SUMMARY:
This study will be done at Ain Shams university maternity hospital to identify the significant risk of maternal intensive care unit admission, need for advanced surgery, postpartum hemorrhage, need for blood transfusion, febrile morbidity, neonatal intensive care unit admission (NICU), need for neonatal intubation and low APGAR scoring in both vaginal and cesarean section .and this will lead us to know if cesarean section rates in our unit is a safe alternative to vaginal delivery and which of both maneuvers will introduce fewer hazards to mother and fetus.

DETAILED DESCRIPTION:
* Type of Study: a cross-sectional study
* Study Setting: Ain Shams maternity hospital
* Study Period: 6 months
* Study Population: in this prospective study, all women who deliver vaginally and by cesarean section at Ain Shams maternity hospital will be included.
* Sampling Method: All of the pregnant women who will deliver vaginally and all of pregnant women who will deliver by cesarean sections in the labor delivery room at Ain Shams University Maternity Hospital on a fixed day and by a fixed team over a period of 6 months
* Sample Size: all pregnant women who will deliver at Ain Shams maternity hospital.
* Inclusion criteria :

  * All of the patients who will deliver vaginally
  * All of the patients who will deliver by cesarean sections.
* Exclusion criteria: no exclusion criteria, all women who will attend for delivery will be included.
* Ethical Considerations: the study objectives will be briefly and clearly described to all participants and an oral consent will be obtained from all patients.
* Study Procedures :

In all selected cases the following will be recorded:

Parameters of maternal morbidity:

1. ICU admission due to the complication of delivery.
2. Need for advanced surgery (int. iliac ligation -hysterectomy -or due to the injury of pelvic organs).
3. Febrile morbidity temp >38C on two or more occasion within 48h of delivery.
4. Postpartum hemorrhage (blood loss 500cc in VD and 1liter in C\S).
5. Wound infection.
6. Late complications e.g. (D.V.T-puerperal sepsis and hematoma).
7. Need for blood transfusion post labor
8. Maternal mortality.

Parameters of fetal morbidity:

1. Intracranial hemorrhage as compilations of delivery.
2. Neonatal ICU admission as compilations of delivery
3. Fracture (Femur, ribs, and humorous)
4. Meconium aspiration.
5. Erb's palsy.
6. APGARscore1-5.
7. Need for intubation during resuscitation.

   * Statistical analysis The patient will be subdivided into 4 groups, normal VD, instrumental VD, emergency C\S, and elective C\S The data has been collected in analytical sheet tabulated and statistical analysis using the following tests

1- T-test. 2- Chi-square test. 3- Fisher exact test

Statistical package :

data analysis will be performed by SPSS 16.0 using descriptive statistics tools, including mean, standard deviation and figures.A t-test will be used to compare mean values of the two groups .P-values, smaller than 0.05, were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All of the patients who will deliver vaginally
* All of the patients who will deliver by cesarean sections.

Exclusion Criteria:

* no exclusion criteria, all women who will attend for delivery will be included.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: all women who delivered vaginally and by cesarean section at Ain Shams maternity hospital will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
labor and delivery outcome | 24 hours
  document maternal and perinatal morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Tamer F Borg, professor, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt